CLINICAL TRIAL: NCT05013515
Title: A Study of Surufatinib Neoadjuvant Therapy for Locally Advanced Primary Saliary Gland Adenocarcinoma：a Single-arm, Prospective,Open Label Study
Brief Title: Efficacy and Safety of Neoadjuvant Surufatinib for Patients With Salivary Gland Carcinomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-HNC101
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Salivary Gland Carcinomas
MeSH Terms: interventions — surufatinib; Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salivary Gland Carcinomas (Experimental): Patients with Salivary Gland Carcinomas were given Surufatinib .
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Patients receive oral Surufatinib at a dose of 300mg/d (once-daily dosing continuously, every 28-day treatment cycle), A total of 2 cycles were performed, and efficacy evaluation was performed at the end of each cycle or was determined to be required by the investigator. If disease progression or unacceptable toxicity occurred during the period, induction therapy was terminated early, and after corresponding treatment, surgical treatment was entered as early as possible.
  Surufatinib treatment was interrupted 4-7 days before surgical treatment to maintain organ function; Note: Postoperative radiotherapy or chemoradiotherapy is permitted after radical surgery at the discretion of the investigator.
  Other Names: radiotherapy or chemoradiotherapy

SUMMARY:
The objective is to investigate the efficacy and safety of Surufatinib Neoadjuvant Therapy for Locally Advanced Primary Saliary Gland Adenocarcinoma.

DETAILED DESCRIPTION:
The purpose of this study was to explore whether the efficacy and survival time of patients with local advanced primary salivary gland adenocarcinoma could be further improved through the treatment of Surufatinib neoadjuvant for local advanced primary salivary gland adenocarcinoma, and to explore the safety and tolerability of this regimen.A Study of Surufatinib Neoadjuvant Therapy for Locally Advanced Primary Saliary Gland Adenocarcinoma：a Single-arm, Prospective,Open Label Study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures;
2. aged between 18 and 75 years are eligible;
3. Male and Female are available；
4. Patients with locally advanced primary salivary gland adenocarcinoma confirmed by pathology or histology (except nasopharyngeal carcinoma);At least one measurable lesion (≥10mm on spiral CT scan, meeting RECIST 1.1 criteria);
5. Patients have not received chemotherapy or radiotherapy, targeted therapy, or surgery for any previous reason;
6. Patients with indications for surgery；
7. Primary TNM stage Ⅲ-ⅣA (T1-2/N1-2/M0 or T3-4A/CN0-2 /M0, AJCC2018);
8. Patients should not be accompanied by any other anticancer therapy;
9. It is not concomitant with long-term treatment (≥3 months) with ≥20mg daily dose of methylprednisolone or equivalent dose of corticosteroids;
10. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
11. Predicted survival ≥12 weeks;
12. Screening laboratory values must meet the following criteria (within past 14 days):

    * neutrophils ≥3.0×109/L ;
    * platelets ≥100×109/L；
    * hemoglobin ≥ 9.0 g/dL;
    * albumin≥3g/dL；
    * total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; Endogenous creatinine clearance >50ml/min (Cockcroft- Gault formula);
13. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Prior treatment with Surufatinib,or other antiangiogenic drugs were used within 6 months;
2. Prior antitumor therapy with chemotherapy, radical radiation therapy ，biological immunotherapy，targeted therapy within 4 weeks.
3. Prior participation in other clinical trials not approved or listed in China within past 4 weeks；
4. Prior major surgery within past 4 weeks (Venous catheterization, puncture and drainage are excluded);
5. International standardized ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN;
6. Clinically significant severe electrolyte abnormality judged by investigator ;
7. Hypertension that is not controlled by the drug, and is defined as: SBP≥140 mmHg and/or DBP≥90 mmHg;
8. Currently suffering from poorly controlled diabetes (after regular treatment, fasting plasma glucose concentration ≥10mmol/L);
9. The patient currently has disease or condition that affects the absorption of the drug, or the patient cannot be administered orally;
10. Digestive tract disease such as gastric and duodenal active ulcer, ulcerative colitis or unresected tumor, or other conditions determined by the investigator that may cause gastrointestinal bleeding and perforation;
11. Evidence of bleeding tendency or history within 3 months, or thromboembolic event (including a stroke event and/or a transient ischemic attack) occurred within 12 month;
12. Cardiovascular disease of significant clinical significance (myocardial infarction, unstable arrhythmia or unstable angina ，Coronary Artery Bypass Grafting within past 6 months,)；
13. Had other malignant tumors in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled);
14. Active or uncontrolled severe infection (≥CTCAE2 infection);
15. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>2000IU/ml);
16. Evidence with active CNS disease or previous brain metastases;
17. The toxicity associated with previous anti-tumor treatment has not recovered to ≤CTCAE1, except for peripheral neurotoxicity and alopecia ≤CTCAE2 caused by oxaliplatin;
18. Pregnant or nursing;
19. Transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony stimulating factor (G-CSF), had been received within 14 days before enrollment;
20. Tumor involving skin and/or pharyngeal mucosa with ulceration;
21. Patients with a history of psychotropic drug abuse and unable to quit or with mental disorders;
22. Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to doubt is not suitable for the use of study drugs in patients with a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or make the patients at high risk.
23. Routine urine indicated that urine protein ≥2+, and the 24-hour urine protein volume >1.0g;
24. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | up to 12 months
  the reduction of the active tumor below an established clinically significant node.
Progression Free Survival (PFS) | up to 36 months
  To assess the efficacy of Neoadjuvant Surufatinib for Patients With Salivary Gland Carcinomas, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Assess the anti-tumor activity:DCR | up to 12 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival time | through study completion, an average of 1 year
  OS was calculated from the date of pharmacy to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ruan, MD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, China